CLINICAL TRIAL: NCT00583778
Title: A Comparison of Levalbuterol Plus Ipratropium With Levalbuterol Alone in the Treatment of Acute Asthma Exacerbation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: MetroHealth Medical Center (Other)
Collaborators: Sumitomo Pharma America, Inc. (Industry)
Responsible Party: Principal Investigator, Rita Cydulka, MD, Emergency medicine physician, MetroHealth Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IRB04-00127
Record Dates: First submitted 2007-12-20; First posted 2007-12-31 (Estimated); Results first posted 2022-05-16 (Actual); Last update posted 2022-05-16 (Actual); Status verified 2022-05

CONDITIONS: Asthma
Keywords: Asthma; Bronchodilators; Levalbuterol; Ipratropium
MeSH Terms: conditions — Asthma | interventions — Ipratropium

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Levalbuterol (Active Comparator): levalbuterol 1.25 mg every 20 minutes for 3 doses plus placebo (saline)
  Interventions: Drug: ipratropium
- Levalbuterol plus ipratropium (Experimental): ipratropium 0.5 mg nebulized every 20 minutes for 3 doses added to levalbuterol 1.25 mg every 20 minutes for 3 doses
  Interventions: Drug: ipratropium

INTERVENTIONS:
Drug: ipratropium — 0.5 mg of ipratropium added to 1.25 mg levalbuterol given every 20 minutes for 3 doses

SUMMARY:
This is a double blind, controlled clinical trail testing whether three doses of 1.25 mg of nebulized levalbuterol in combination with three doses of 0.5mg of nebulized ipratropium will lead to greater bronchodilation than that achieved by three doses of nebulized 1.25 mg of levalbuterol alone every 20 minutes.

The primary hypothesis of this study is that three doses of 1.25 mg of nebulized levalbuterol in combination with three doses of 0.5mg of nebulized ipratropium will lead to greater bronchodilation than that achieved by three doses of nebulized 1.25 mg of levalbuterol alone every 20 minutes. The secondary hypothesis is that the treatment combination of levalbuterol and ipratropium will lead to fewer hospitalizations than levalbuterol alone in patients with acute asthma exacerbation. Other secondary objectives include (1) evaluating the relationship between baseline (S)- albuterol levels and (R)- albuterol levels on presentation and FEV1, (2) the relationship between baseline (S)- albuterol levels and (R)- albuterol levels on presentation and change in FEV1,(3) time to event analysis for an improvement of 15%, 20%, 30%, 40%, and 50% in FEV1 from initial presentation value, (4) analysis of FEV1 at discharge.

DETAILED DESCRIPTION:
Patients will then receive, in a randomized double-blinded fashion, levalbuterol, 1.25mg every 20 minutes for a total of 3 aerosolized doses combined with ipratropium, 0.5mg every 20 minutes for a total of 3 aerosolized doses. The medication will be premixed by the pharmacy in a total of 3 ml of normal saline and the nebulizer will be driven with oxygen at 6 liters per minute. A second plasma sample for analysis of albuterol isomers will be drawn within a fifteen minute window following the third aerosol treatment. Spirometry will be repeated again at 30 and 60 minutes after the third aerosol treatment (Figure 1). All patients will receive prednisone, 60mg orally immediately after their first dose of aerosolized medications, unless contraindications to prednisone administration are present. Patients will not receive any other medications during the time course of the study. Vital signs and pulse oximetry will be repeated prior to each nebulized treatment and again 30 minutes after the third nebulized treatment.

The study will terminate 60 minutes after the third aerosol administration. At that point, any further therapy will be at the discretion of the treating physician. Patients will be questioned about the occurrence of any side effects from levalbuterol treatment including palpitations, anxiety, nausea, vomiting or headache. Patients will also be questioned about the occurrence of any side effects from ipratropium, including dry mouth, dry eyes, and urinary retention. Patients will be withdrawn from the study at any point these side effects become intolerable to the patient or any time the patient so desires. Patients will also be withdrawn if they develop palpitations and have an ECG that demonstrates ventricular or supraventricular tachycardia.

.Patients will be called 14 days after their ED visit to assess relapse or recurrence of acute asthma exacerbation. In addition, a chart review will be performed to assess relapse or recurrence of acute asthma exacerbation, as well as determine hospital length of stay in those patients who required admission after the initial visit.

ELIGIBILITY:
Inclusion Criteria:

* 18-45 years of age
* history of asthma
* FEV1 > 50% of predicted for their height, age, gender and race upon presentation to the ED
* no other cause of wheezing or shortness of breath except for asthma as determined by the Investigator
* no history of glaucoma
* no Ipratropium or other anticholinergics within 6 hours of study

Exclusion Criteria:

* subjects who, in the investigator's opinion, have life-threatening asthma requiring emergent intervention precluding the ability to complete the treatments during the treatment period
* based upon history or physical exam in the ED orClinic, subjects with known or suspected cause of pulmonary symptoms other than asthma, such as COPD, CHF, pneumonia, pulmonary embolism, or angioedema
* subject with a known sensitivity to levalbuterol or racemic albuterol
* known 20 pack year smoker
* use of ipratropium 6 hours prior to presenting to the ED
* subject who may be pregnant or is pregnant es evidenced by pregnancy test

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 141 (Actual)
Dates: Start 2004-08; Primary Completion 2008-11 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rita K Cydulkla, MD, Principal Investigator — MetroHealth Medical Center
Locations (1):
- MetroHealth Medical Center, Cleveland, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Adult patients between the ages if 18 and 45 years presenting to the emergency department with acute asthma. They were enrolled by one of the study nurses. Patients were eligible to enroll if their FEV-1 was less than 50% predicted on arrival. Enrollment occurred between December 2005 and December 2008.
Period: Overall Study
Arm/Group | Levalbuterol | Levalbuterol Plus Ipratropium
Started | 74 | 67
Completed | 74 | 67
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Levalbuterol | Levalbuterol Plus Ipratropium | Total
Number analyzed (Participants) | 74 | 67 | 141
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 74 | 67 | 141
  >=65 years | 0 | 0 | 0
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 31.1 [24 to 38] | 30.3 [23 to 37] | 30.6 [24 to 37]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 54 | 36 | 90
  Male | 20 | 31 | 51
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 74 | 67 | 141

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Bronchodilation
Description: Measure FEV-1 in participants immediately prior to treatment and 60 minutes after final treatment to determine improvement in bronchodilation after 1.25mg nebulized levalbuterol + 0.5mg nebulized ipratropium administered every 20 minutes for a total of 3 doses versus bronchodilation after 1.25mg nebulized levalbuterol administered every 20 minutes for a total of 3 doses. FEV-1 measurements were obtained using a hand held spirometer. A difference in 12% of median FEV-1 measures between the two groups was considered clinically significant. Patients were called 14 days after their ED visit to assess relapse or recurrence of acute asthma exacerbation. In addition, a chart review was performed to assess relapse or recurrence of acute asthma exacerbation, as well as determine hospital length of stay in those patients who required admission after the initial visit.
Time Frame: FEV-1 measured Immediately before treatment dose 1 & 60 minutes after completion of treatment dose 3. Assessment of relapse or recurrence were determined at day 14 after the ED visit.
Measure: Count of Participants; unit: Participants
Arm/Group | Levalbuterol | Levalbuterol Plus Ipratropium
Number analyzed (Participants) | 141 | 141
Participants | 74 | 67

2. Primary Outcome: Change in FEV-1 % Predicted Over Time
Description: Primary Outcome- the difference in FEV-1at 60 minutes between participants who received Levalbuterol 1.25 mg x 3 vs participants who received Levalbuterol 1.25 mg x3 + Ipratropium 0.5 mg x3
Time Frame: 60 minutes
Population: Overall Number of Participants Analyzed 141
Measure: Median (Inter-Quartile Range); unit: percentage of FEV-1 predicted
Arm/Group | Levalbuterol | Levalbuterol Plus Ipratropium
Number analyzed (Participants) | 74 | 67
percentage of FEV-1 predicted | 45 [37 to 58] | 47 [40 to 63]
Statistical Analysis 1: Comparison: Levalbuterol vs Levalbuterol Plus Ipratropium; Data were analyzed using STATA 10 SE.Categorical variables were described using frequencies and relative frequencies. Distribution of continuous variables were evaluated for normality using the Shapiro-Walk test and graphically using histograms and box plots. Because most data were non-parametric, they were described using the median and 25th and 75th percentiles (interquartile range) and then compared using Wilcoxon rank sum test; Test type: Superiority; p < 0.05, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = 12, Standard Deviation 25; This study was designed to detect an absolute difference of 12 % in change of FEV-1percent predicted, with a standard deviation of 25% based on data provided to us from previous studies conducted by Sepracor. Based on this assumption, we sought to enter 76 patients in each group to have an 80% power to detect a 12 % absolute difference in charge of FEV-1 percent predicted over time at an alpha of 0.05. This accounted for a potential 10% dropout rate after randomization

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Levalbuterol | Levalbuterol Plus Ipratropium
All-Cause Mortality (participants affected / at risk) | 0/74 | 0/67
Serious Adverse Events (participants affected / at risk) | 0/74 | 0/67
Other Adverse Events (participants affected / at risk) | 0/74 | 0/67

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No